CLINICAL TRIAL: NCT00570011
Title: Efficacy of Two Different Dose Regimens of Somatropin in Growth Hormone Deficient Adult Patients
Brief Title: Low and Conventional Dose of Somatropin in Growth Hormone Deficient Adult Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: University of Naples (Other); University of Padova (Other); University of Milan (Other); University of Pisa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 822; B9R-EW-GDED
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Last update posted 2007-12-11 (Estimated); Status verified 2007-12

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Somatropin
- 2 (Experimental)
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — 3 microg/kg/day for the first three months.The dose was then doubled (6 microg/kg/day) for the next three-months.
  Other Names: LLY137998
  Arms: 1
Drug: Somatropin — 6 microg/kg/day for the first three months. The dose was then doubled (12 microg/kg/day) for the next three-months.
  Other Names: LLY137998
  Arms: 2

SUMMARY:
An international study in which patients with GHD were randomized to receive somatropin at a dose of either 3 microg/kg/day or 6 microg/kg/day for the first three months. The dose was then doubled (6 microg/kg/day, LD or 12 microg/kg/day, CD) for the next three-months.

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study only if they meet all of the following criteria:

1. Adult males and females with GHD, arising during adult life from pituitary ablation or failure, onset of GHD have taken place at least 1 year before entering the study, or,
2. Adult males and females with GHD either idiopathic or secondary to pituitary disease arising in childhood.
3. Demonstrated GHD as documented by a negative response to a standard GH stimulation test within the last 5 years previous year (see Section 3.4.3, part b). Maximal peak must be less than 3.0 ng/ml.
4. Receiving replacement for other deficient hormones for at least 3 months prior to the start of the study, where necessary.
5. Have given informed consent.

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

1. Patients with clinically significant pulmonary, cardiac, hepatic, renal or neuromuscular disease or with chromosomal or genetic malformation syndromes.
2. Patients who have any evidence of an active tumorous process. Intercranial lesions must be inactive and any antitumour therapy must be complete.
3. Pregnant women and lactating females or women who decide to become pregnant during the study and who are not taking adequate contraceptives.
4. Patients thought unlikely to comply with the protocol.
5. Patients taking an investigational drug in the previous month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 1997-06; Study Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Plasminogen activator inhibitor-1 (PAI-1) and tissue plasminogen activator (t-PA) as a function of changes in insulin levels was investigated. | 6 months

SECONDARY OUTCOMES:
Serum concentrations of Leptin, Insulin, IGFBP1, IGFBP2, IGF2 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com